CLINICAL TRIAL: NCT04107532
Title: Cognitive Behavioral Therapy Based on Virtual Reality and Biofeedback Technology
Acronym: VRET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chun Wang, associate chief physician, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-KY095
Record Dates: First submitted 2019-09-04; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Virtual Reality Exposure Therapy
MeSH Terms: interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Therapy for Acrophobia (Other): There were a total of 5 treatments in the VR treatment group, followed by cliffs, cliffs, cliffs, single-plank bridges, and high-altitude rescues. The difficulty of the scene increased in turn. The frequency of treatment twice a week, about 30 minutes each time, fills in the motion sickness questionnaire before and after each treatment to understand the safety of VR treatment. In the course of treatment, physiological data such as skin electricity, skin temperature, heart rate, and blood volume were measured, and the state of the subjects was objectively evaluated. At the same time, every two minutes, participants were asked about sud values and recorded.
  Interventions: Other: Virtual Reality Therapy and Imagination Exposure Therapy
- Imagination Exposure Therapy for Acrophobia (Other): The imaginary exposure treatment program is to convert the five scenes of VR exposure treatment through language, guide the subjects through the guidance language, guide the subjects to expose, and achieve the purpose of adaptation. Both treatment groups were required to collect scales and nuclear magnetic data before, after and after six months of follow-up.
  Interventions: Other: Virtual Reality Therapy and Imagination Exposure Therapy

INTERVENTIONS:
Other: Virtual Reality Therapy and Imagination Exposure Therapy — Virtual Reality Therapy and Imagination Exposure Therapy

SUMMARY:
The subjects were randomly assigned to VR treatment group and imaginary leak treatment group. In the VR treatment group, there were six VR exposure experiences, ranging from low to high levels of exposure, about 20 minutes each time, twice a week. During the course of treatment, physiological data such as skin electricity, skin temperature, heart rate and blood volume were measured, and the state of the subjects was evaluated more objectively. At the same time, every two minutes, the participants were asked the SUD value and recorded. AQ, ATHQ and BAT were recorded before treatment, after treatment and during the follow-up period of six months. The two groups were treated differently. n addition, at the beginning of this treatment program, an experimental study was added to understand the eye movement characteristics of patients with acrophobia. By viewing a group of high-altitude pictures, recording their eye movement characteristics and physiological feedback data, and scoring the anxiety level of each picture, and joining the normal control group, we can find a group of high-altitude pictures which can cause high-altitude fear in patients with high-altitude fear, and lay a foundation for future related research.

DETAILED DESCRIPTION:
The study recruited 60 patients with Acrophobia and randomly assigned them to the VR treatment group and the imaginary exposure treatment group. Recruitment conditions for Acrophobia: The Acrophobia questionnaire scored more than 45.45 points; Age 18-55 years old; Right-handedness; No psychotherapy or psychiatric medication for six months; Normal vision or corrective vision; Not during pregnancy or lactation. Before the formal treatment, the participants were interviewed, mainly to understand in detail the fear of heights in the subjects, and to tell the subjects the reasons for the fear of heights and the principles of our treatment. After confirming the participants 'intention to participate in the treatment, a heart test was conducted to eliminate heart problems and finally sign an informed consent form. At the end of the interview, pre-tests were performed to collect fear of heights questionnaires, high attitude questionnaires, behavioral avoidance tests, and nuclear magnetic data collection. There were a total of 5 treatments in the VR treatment group, followed by cliffs, cliffs, cliffs, single-plank bridges, and high-altitude rescues. The difficulty of the scene increased in turn. The frequency of treatment twice a week, about 30 minutes each time, fills in the motion sickness questionnaire before and after each treatment to understand the safety of VR treatment. In the course of treatment, physiological data such as skin electricity, skin temperature, heart rate, and blood volume were measured, and the state of the subjects was objectively evaluated. At the same time, every two minutes, participants were asked about sud values and recorded. Visualizing exposure therapy is to achieve the goal of exposure by transforming the five scenes of VR exposure therapy through language and guiding the subjects through the guidance language. Both treatment groups were required to collect scales and nuclear magnetic data before, after and after six months of follow-up. In addition, at the beginning of this treatment program, an experimental study was added to understand the characteristics of eye movement in people with anorexia. By looking at high altitude images, recording their eye movement characteristics and physiological feedback, and rating the anxiety levels of each image, adding to the normal control group, we found a high altitude image that can cause high altitude fear in people with high altitude fear. And lay the foundation for future related research.

ELIGIBILITY:
Inclusion Criteria:

1.18-55 years old; 2.The anxiety scale in AQ scored more than 45.45 points ; 3.Meeting the DSM-IV criteria for specific phobia.

Exclusion Criteria:

1. Other current or recent mental disorders, such as post-traumatic stress disorder;
2. Other physical diseases (such as heart disease and epilepsy) that may affect treatment;
3. Pregnancy or lactation;
4. No effect of psychotropic drugs or psychotherapy or prior exposure to heightphobia within 6 months (2013).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
AQ | 3 weeks
  There were a total of 20 questions on the anxiety scale in the Acrophobia Questionnaire. Each topic scored 0-6 points. More than 45.45 points were included in the group to assess the differences in scores between the subjects before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Chun Wang, doc., Study Chair — Nanjing Brain Hospital Nanjing, Jiangsu China

IPD SHARING:
Plan to Share IPD: Undecided